CLINICAL TRIAL: NCT02547571
Title: The Bowel CLEAnsing: A National Initiative
Acronym: B-CLEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alan Barkun (Other)
Collaborators: Pendopharm (Industry)
Responsible Party: Sponsor-Investigator, Alan Barkun, Gatroenterologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V2015-001
Record Dates: First submitted 2015-09-01; First posted 2015-09-11 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Subjets Requiring a Colonoscopy
Keywords: Outpatient
MeSH Terms: interventions — Golytely

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- 1) Early colonoscopy; 2) High-dose, split-dose; 3)Clear liquid (Active Comparator)
  Interventions: Drug: High volume PEG split-dose; Other: Clear liquid diet; Other: Early colonoscopy (stratified)
- 1) Early colonoscopy; 2) High-dose, split-dose; 3)Low residue (Active Comparator)
  Interventions: Drug: High volume PEG split-dose; Other: Low residue diet; Other: Early colonoscopy (stratified)
- 1) Early colonoscopy; 2) Low volume split-dose; 3)Clear liquid (Active Comparator)
  Interventions: Drug: Low volume PEG split-dose; Other: Clear liquid diet; Other: Early colonoscopy (stratified)
- 1) Early colonoscopy; 2) Low volume split-dose; 3)Low residue (Active Comparator)
  Interventions: Drug: Low volume PEG split-dose; Other: Low residue diet; Other: Early colonoscopy (stratified)
- 1) Early colonoscopy; 2) High-dose, day before; 3)Clear liquid (Active Comparator)
  Interventions: Drug: High volume PEG non split, day before; Other: Clear liquid diet; Other: Early colonoscopy (stratified)
- 1) Early colonoscopy; 2) High-dose, day before; 3)Low residue (Active Comparator)
  Interventions: Drug: High volume PEG non split, day before; Other: Low residue diet; Other: Early colonoscopy (stratified)
- 1) Later colonoscopy; 2) High-dose, split-dose; 3)Clear liquid (Active Comparator)
  Interventions: Drug: High volume PEG split-dose; Other: Clear liquid diet; Other: Later colonoscopy (stratified)
- 1) Later colonoscopy; 2) High-dose, split-dose; 3)Low residue (Active Comparator)
  Interventions: Drug: High volume PEG split-dose; Other: Low residue diet; Other: Later colonoscopy (stratified)
- 1) Later colonoscopy; 2) Low volume split-dose; 3)Clear liquid (Active Comparator)
  Interventions: Drug: Low volume PEG split-dose; Other: Clear liquid diet; Other: Later colonoscopy (stratified)
- 1) Later colonoscopy; 2) Low volume split-dose; 3)Low residue (Active Comparator)
  Interventions: Drug: Low volume PEG split-dose; Other: Low residue diet; Other: Later colonoscopy (stratified)
- 1) Later colonoscopy; 2) Low volume day before; 3)Clear liquid (Active Comparator)
  Interventions: Drug: Low volume PEG non split, same day; Other: Clear liquid diet; Other: Later colonoscopy (stratified)
- 1) Later colonoscopy; 2) Low volume day before; 3)Low residue (Active Comparator)
  Interventions: Drug: Low volume PEG non split, same day; Other: Low residue diet; Other: Later colonoscopy (stratified)

INTERVENTIONS:
Drug: High volume PEG split-dose — Colyte® or PegLyte® will be provided to the subject who will be asked to drink 2L of the preparation starting at 7:00 PM the day before the procedure at a rate of 240 mL every 10 minutes until completed. The second dose of 2L of preparation will be taken the morning of the colonoscopy starting 4-5 hours prior to the planned procedural time at a rate of 240 mL every 10 minutes until completed.
  Other Names: Colyte® or PegLyte®
  Arms: 1) Early colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Early colonoscopy; 2) High-dose, split-dose; 3)Low residue; 1) Later colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) High-dose, split-dose; 3)Low residue
Drug: Low volume PEG split-dose — Bi-PegLyte® will be provided to the subject who will be asked to ingest 3 tabs of Bisacodyl 5 mg (total 15 mg) at 2:00 PM the day before the procedure. After the first bowel movement, or if there is no bowel movement within 6 hours of taking the Bisacodyl tablets, the subject will be asked to drink 1L of the solution at a rate of 240 mL every 10 minutes until the solution is completed. The second dose of 1L of preparation will be taken the morning of the colonoscopy starting 4-5 hours prior to the procedure at a rate of 240 mL every 10 minutes. Use of antacids will not be permitted within one hour of taking bisacodyl.
  Other Names: Bi-PegLyte®
  Arms: 1) Early colonoscopy; 2) Low volume split-dose; 3)Clear liquid; 1) Early colonoscopy; 2) Low volume split-dose; 3)Low residue; 1) Later colonoscopy; 2) Low volume split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume split-dose; 3)Low residue
Drug: High volume PEG non split, day before — Colyte® or PegLyte® will be provided to the subject who will be asked to drink 4L of preparation starting at 6:00 PM the day before the procedure, at a rate of 240 mL every 10 minutes until completed.
  Other Names: Colyte® or PegLyte®
  Arms: 1) Early colonoscopy; 2) High-dose, day before; 3)Clear liquid; 1) Early colonoscopy; 2) High-dose, day before; 3)Low residue
Drug: Low volume PEG non split, same day — Bi-PegLyte® will be provided to the subject, who will be asked to ingest 3 tabs of Bisacodyl 5 mg (total 15 mg) at 2:00 PM the day before the procedure and will drink 2L of preparation the morning of the colonoscopy starting 4 hours prior to the procedure at a rate of 240 mL every 10 minutes, until completed. Use of antacids will not be permitted within one hour of taking Bisacodyl.
  Other Names: Bi-PegLyte®
  Arms: 1) Later colonoscopy; 2) Low volume day before; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume day before; 3)Low residue
Other: Clear liquid diet
  Arms: 1) Early colonoscopy; 2) High-dose, day before; 3)Clear liquid; 1) Early colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Early colonoscopy; 2) Low volume split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume day before; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume split-dose; 3)Clear liquid
Other: Low residue diet
  Arms: 1) Early colonoscopy; 2) High-dose, day before; 3)Low residue; 1) Early colonoscopy; 2) High-dose, split-dose; 3)Low residue; 1) Early colonoscopy; 2) Low volume split-dose; 3)Low residue; 1) Later colonoscopy; 2) High-dose, split-dose; 3)Low residue; 1) Later colonoscopy; 2) Low volume day before; 3)Low residue; 1) Later colonoscopy; 2) Low volume split-dose; 3)Low residue
Other: Early colonoscopy (stratified) — "Early" appointments: 7:30 AM to 10h30 AM
  Arms: 1) Early colonoscopy; 2) High-dose, day before; 3)Clear liquid; 1) Early colonoscopy; 2) High-dose, day before; 3)Low residue; 1) Early colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Early colonoscopy; 2) High-dose, split-dose; 3)Low residue; 1) Early colonoscopy; 2) Low volume split-dose; 3)Clear liquid; 1) Early colonoscopy; 2) Low volume split-dose; 3)Low residue
Other: Later colonoscopy (stratified) — "Later" appointments: 10:30 AM to 4:30 PM.
  Arms: 1) Later colonoscopy; 2) High-dose, split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) High-dose, split-dose; 3)Low residue; 1) Later colonoscopy; 2) Low volume day before; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume day before; 3)Low residue; 1) Later colonoscopy; 2) Low volume split-dose; 3)Clear liquid; 1) Later colonoscopy; 2) Low volume split-dose; 3)Low residue

SUMMARY:
The purpose of this study is to compare diet, type of bowel preparation and time of colonoscopy to determine if one method is better than the other and, if they are the same, identify the one which is the most convenient for the patients.

DETAILED DESCRIPTION:
The objective of the current proposed trial is thus to compare the cleanliness achieved with PEG high-volume (2L+2L) split-dose versus PEG (1L+1L)+Bisacodyl low-volume split-dose, or PEG high volume (4L) non-split day before versus PEG low volume (2L) non-split same day preparation, according to time of endoscopy (early or later), as well as assess the role of diet (low residue or clear liquid diet) according to these different Canadian outpatient preparation regimens.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* 18 years or older
* Able to comprehend the trial
* Have an indication for full colonoscopy

Exclusion Criteria:

Subjects are excluded from enrollment into the study if any of the following are present:

General exclusion criteria:

* Subject refusal
* Previous bowel preparation in the last 14 days
* Pregnancy or breastfeeding
* Reduced mobility

Medical/Endoscopic exclusion criteria:

* Suspected or diagnosed with bowel obstruction
* Any colonic surgery
* Toxic megacolon
* Ileus
* Ischemic colitis
* Decompensated heart failure
* Severe acute renal failure
* Severe liver disease
* Severe electrolyte imbalance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3476 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing according to the Boston Scale | Day of colonoscopy

SECONDARY OUTCOMES:
Subject willingness to repeat the preparation (survey) | Day of colonoscopy
Withdrawal time and total procedural time | Day of colonoscopy
Cecal or ileal intubation rate for colonoscopies | Day of colonoscopy
Polyp detection and polypectomy rate | Day of colonoscopy
Right colon polyp detection rate | Day of colonoscopy
Specific lesional rates identified according to pathology | up to 30 days
% of preparation taken by the subject | Day of colonoscopy
Subject travel time to endoscopy unit (hrs) | Day of colonoscopy
Incontinence | Day of colonoscopy
Fecal Immunochemical Test value | Day of colonoscopy
Montreal score compared to BBPS | Day of colonoscopy
Ottawa Bowel Preparation Scores compared to BBPS | Day of colonoscopy

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (10):
  - Forzani & MacPhail Colon Cancer Screening Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences center and St. Boniface Hospital, Winnipeg, Manitoba
  - QEII HSC, Halifax, Nova Scotia
  - Western University, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - CHUM, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital St-Sacrement, CHU de Québec-Université Laval, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Assal C, Watson PY. Angioedema as a hypersensitivity reaction to polyethylene glycol oral electrolyte solution. Gastrointest Endosc. 2006 Aug;64(2):294-5. doi: 10.1016/j.gie.2006.02.008. Epub 2006 May 19. No abstract available. PMID 16860094
- [Result] Brahmania M, Ou G, Bressler B, Ko HK, Lam E, Telford J, Enns R. 2 L versus 4 L of PEG3350 + electrolytes for outpatient colonic preparation: a randomized, controlled trial. Gastrointest Endosc. 2014 Mar;79(3):408-416.e4. doi: 10.1016/j.gie.2013.08.035. Epub 2013 Oct 24. PMID 24206747
- [Result] Bucci C, Rotondano G, Hassan C, Rea M, Bianco MA, Cipolletta L, Ciacci C, Marmo R. Optimal bowel cleansing for colonoscopy: split the dose! A series of meta-analyses of controlled studies. Gastrointest Endosc. 2014 Oct;80(4):566-576.e2. doi: 10.1016/j.gie.2014.05.320. Epub 2014 Jul 19. PMID 25053529
- [Result] Cesaro P, Hassan C, Spada C, Petruzziello L, Vitale G, Costamagna G. A new low-volume isosmotic polyethylene glycol solution plus bisacodyl versus split-dose 4 L polyethylene glycol for bowel cleansing prior to colonoscopy: a randomised controlled trial. Dig Liver Dis. 2013 Jan;45(1):23-7. doi: 10.1016/j.dld.2012.07.011. Epub 2012 Aug 21. PMID 22917636
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Chorev N, Chadad B, Segal N, Shemesh I, Mor M, Plaut S, Fraser G, Geller A, Gal E, Niv Y. Preparation for colonoscopy in hospitalized patients. Dig Dis Sci. 2007 Mar;52(3):835-9. doi: 10.1007/s10620-006-9591-5. PMID 17253131
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Result] de Leone A, Tamayo D, Fiori G, Ravizza D, Trovato C, De Roberto G, Fazzini L, Dal Fante M, Crosta C. Same-day 2-L PEG-citrate-simethicone plus bisacodyl vs split 4-L PEG: Bowel cleansing for late-morning colonoscopy. World J Gastrointest Endosc. 2013 Sep 16;5(9):433-9. doi: 10.4253/wjge.v5.i9.433. PMID 24044042
- [Result] El Sayed AM, Kanafani ZA, Mourad FH, Soweid AM, Barada KA, Adorian CS, Nasreddine WA, Sharara AI. A randomized single-blind trial of whole versus split-dose polyethylene glycol-electrolyte solution for colonoscopy preparation. Gastrointest Endosc. 2003 Jul;58(1):36-40. doi: 10.1067/mge.2003.318. PMID 12838218
- [Result] Eun CS, Han DS, Hyun YS, Bae JH, Park HS, Kim TY, Jeon YC, Sohn JH. The timing of bowel preparation is more important than the timing of colonoscopy in determining the quality of bowel cleansing. Dig Dis Sci. 2011 Feb;56(2):539-44. doi: 10.1007/s10620-010-1457-1. Epub 2010 Nov 2. PMID 21042853
- [Result] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Result] Hangartner PJ, Munch R, Meier J, Ammann R, Buhler H. Comparison of three colon cleansing methods: evaluation of a randomized clinical trial with 300 ambulatory patients. Endoscopy. 1989 Nov;21(6):272-5. doi: 10.1055/s-2007-1012967. PMID 2693078
- [Result] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Result] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Result] Hendry PO, Jenkins JT, Diament RH. The impact of poor bowel preparation on colonoscopy: a prospective single centre study of 10,571 colonoscopies. Colorectal Dis. 2007 Oct;9(8):745-8. doi: 10.1111/j.1463-1318.2007.01220.x. Epub 2007 Mar 7. PMID 17477852
- [Result] Jayanthi V, Ramathilakam B, Malathi S, Dinakaran N, Balasubramanian V. Comparison of polyethylene glycol versus combination of magnesium sulphate and bisacodyl for colon preparation. Trop Gastroenterol. 2000 Jan-Mar;21(1):18-9. PMID 10835955
- [Result] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Result] Jung YS, Seok HS, Park DI, Song CS, Kim SE, Lee SH, Eun CS, Han DS, Kim YS, Lee CK. A clear liquid diet is not mandatory for polyethylene glycol-based bowel preparation for afternoon colonoscopy in healthy outpatients. Gut Liver. 2013 Nov;7(6):681-7. doi: 10.5009/gnl.2013.7.6.681. Epub 2013 Aug 14. PMID 24312709
- [Result] Khan MA, Piotrowski Z, Brown MD. Patient acceptance, convenience, and efficacy of single-dose versus split-dose colonoscopy bowel preparation. J Clin Gastroenterol. 2010 Apr;44(4):310-1. doi: 10.1097/MCG.0b013e3181c2c92a. No abstract available. PMID 19935082
- [Result] Ko CW, Dominitz JA. Complications of colonoscopy: magnitude and management. Gastrointest Endosc Clin N Am. 2010 Oct;20(4):659-71. doi: 10.1016/j.giec.2010.07.005. PMID 20889070
- [Result] Lawrance IC, Willert RP, Murray K. A validated bowel-preparation tolerability questionnaire and assessment of three commonly used bowel-cleansing agents. Dig Dis Sci. 2013 Apr;58(4):926-35. doi: 10.1007/s10620-012-2449-0. Epub 2012 Oct 25. PMID 23095990
- [Result] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Result] Manno M, Pigo F, Manta R, Barbera C, Bertani H, Mirante VG, Dabizzi E, Caruso A, Olivetti G, Hassan C, Zullo A, Conigliaro R. Bowel preparation with polyethylene glycol electrolyte solution: optimizing the splitting regimen. Dig Liver Dis. 2012 Jul;44(7):576-9. doi: 10.1016/j.dld.2012.02.012. Epub 2012 Mar 26. PMID 22456624
- [Result] Marmo R, Rotondano G, Riccio G, Marone A, Bianco MA, Stroppa I, Caruso A, Pandolfo N, Sansone S, Gregorio E, D'Alvano G, Procaccio N, Capo P, Marmo C, Cipolletta L. Effective bowel cleansing before colonoscopy: a randomized study of split-dosage versus non-split dosage regimens of high-volume versus low-volume polyethylene glycol solutions. Gastrointest Endosc. 2010 Aug;72(2):313-20. doi: 10.1016/j.gie.2010.02.048. Epub 2010 Jun 19. PMID 20561621
- [Result] Martel M, Barkun AN, Menard C, Restellini S, Kherad O, Vanasse A. Split-Dose Preparations Are Superior to Day-Before Bowel Cleansing Regimens: A Meta-analysis. Gastroenterology. 2015 Jul;149(1):79-88. doi: 10.1053/j.gastro.2015.04.004. Epub 2015 Apr 8. PMID 25863216
- [Result] Matro R, Shnitser A, Spodik M, Daskalakis C, Katz L, Murtha A, Kastenberg D. Efficacy of morning-only compared with split-dose polyethylene glycol electrolyte solution for afternoon colonoscopy: a randomized controlled single-blind study. Am J Gastroenterol. 2010 Sep;105(9):1954-61. doi: 10.1038/ajg.2010.160. Epub 2010 Apr 20. PMID 20407434
- [Result] Parente F, Marino B, Crosta C. Bowel preparation before colonoscopy in the era of mass screening for colo-rectal cancer: a practical approach. Dig Liver Dis. 2009 Feb;41(2):87-95. doi: 10.1016/j.dld.2008.06.005. Epub 2008 Jul 26. PMID 18676211
- [Result] Park DI, Park SH, Lee SK, Baek YH, Han DS, Eun CS, Kim WH, Byeon JS, Yang SK. Efficacy of prepackaged, low residual test meals with 4L polyethylene glycol versus a clear liquid diet with 4L polyethylene glycol bowel preparation: a randomized trial. J Gastroenterol Hepatol. 2009 Jun;24(6):988-91. doi: 10.1111/j.1440-1746.2009.05860.x. PMID 19638081
- [Result] Park SS, Sinn DH, Kim YH, Lim YJ, Sun Y, Lee JH, Kim JY, Chang DK, Son HJ, Rhee PL, Rhee JC, Kim JJ. Efficacy and tolerability of split-dose magnesium citrate: low-volume (2 liters) polyethylene glycol vs. single- or split-dose polyethylene glycol bowel preparation for morning colonoscopy. Am J Gastroenterol. 2010 Jun;105(6):1319-26. doi: 10.1038/ajg.2010.79. Epub 2010 May 18. PMID 20485282
- [Result] Parra-Blanco A, Nicolas-Perez D, Gimeno-Garcia A, Grosso B, Jimenez A, Ortega J, Quintero E. The timing of bowel preparation before colonoscopy determines the quality of cleansing, and is a significant factor contributing to the detection of flat lesions: a randomized study. World J Gastroenterol. 2006 Oct 14;12(38):6161-6. doi: 10.3748/wjg.v12.i38.6161. PMID 17036388
- [Result] Rabeneck L, Saskin R, Paszat LF. Onset and clinical course of bleeding and perforation after outpatient colonoscopy: a population-based study. Gastrointest Endosc. 2011 Mar;73(3):520-3. doi: 10.1016/j.gie.2010.10.034. Epub 2010 Dec 31. PMID 21195406
- [Result] Rex DK, Bond JH, Winawer S, Levin TR, Burt RW, Johnson DA, Kirk LM, Litlin S, Lieberman DA, Waye JD, Church J, Marshall JB, Riddell RH; U.S. Multi-Society Task Force on Colorectal Cancer. Quality in the technical performance of colonoscopy and the continuous quality improvement process for colonoscopy: recommendations of the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2002 Jun;97(6):1296-308. doi: 10.1111/j.1572-0241.2002.05812.x. No abstract available. PMID 12094842
- [Result] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Result] Schuman E, Balsam PE. Probable anaphylactic reaction to polyethylene glycol electrolyte lavage solution. Gastrointest Endosc. 1991 May-Jun;37(3):411. doi: 10.1016/s0016-5107(91)70761-x. No abstract available. PMID 2071010
- [Result] Scott SR, Raymond PL, Thompson WO, Galt DJ. Efficacy and tolerance of sodium phosphates oral solution after diet liberalization. Gastroenterol Nurs. 2005 Mar-Apr;28(2):133-9. doi: 10.1097/00001610-200503000-00008. PMID 15832114
- [Result] Seo EH, Kim TO, Park MJ, Heo NY, Park J, Yang SY. Low-volume morning-only polyethylene glycol with specially designed test meals versus standard-volume split-dose polyethylene glycol with standard diet for colonoscopy: a prospective, randomized trial. Digestion. 2013;88(2):110-8. doi: 10.1159/000353244. Epub 2013 Aug 15. PMID 23949563
- [Result] Shah S, Prematta T, Adkinson NF, Ishmael FT. Hypersensitivity to polyethylene glycols. J Clin Pharmacol. 2013 Mar;53(3):352-5. doi: 10.1177/0091270012447122. Epub 2013 Jan 24. No abstract available. PMID 23444288
- [Result] Sharma VK, Nguyen CC, Crowell MD, Lieberman DA, de Garmo P, Fleischer DE. A national study of cardiopulmonary unplanned events after GI endoscopy. Gastrointest Endosc. 2007 Jul;66(1):27-34. doi: 10.1016/j.gie.2006.12.040. PMID 17591470
- [Result] Siddique S, Lopez KT, Hinds AM, Ahmad DS, Nguyen DL, Matteson-Kome ML, Puli SR, Bechtold ML. Miralax with gatorade for bowel preparation: a meta-analysis of randomized controlled trials. Am J Gastroenterol. 2014 Oct;109(10):1566-74. doi: 10.1038/ajg.2014.238. Epub 2014 Aug 19. PMID 25135007
- [Result] Siddiqui AA, Yang K, Spechler SJ, Cryer B, Davila R, Cipher D, Harford WV. Duration of the interval between the completion of bowel preparation and the start of colonoscopy predicts bowel-preparation quality. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):700-6. doi: 10.1016/j.gie.2008.09.047. PMID 19251013
- [Result] Soweid AM, Kobeissy AA, Jamali FR, El-Tarchichi M, Skoury A, Abdul-Baki H, El-Zahabi L, El-Sayyed A, Barada KA, Sharara AI, Mourad F, Arabi A. A randomized single-blind trial of standard diet versus fiber-free diet with polyethylene glycol electrolyte solution for colonoscopy preparation. Endoscopy. 2010 Aug;42(8):633-8. doi: 10.1055/s-0029-1244236. Epub 2010 Jul 9. PMID 20623443
- [Result] Stollman N, Manten HD. Angioedema from oral polyethylene glycol electrolyte lavage solution. Gastrointest Endosc. 1996 Aug;44(2):209-10. doi: 10.1016/s0016-5107(96)70150-5. No abstract available. PMID 8858338
- [Result] Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE; American Society of Colon and Rectal Surgeons; American Society for Gastrointestinal Endoscopy; Society of American Gastrointestinal and Endoscopic Surgeons. A consensus document on bowel preparation before colonoscopy: prepared by a task force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Gastrointest Endosc. 2006 Jun;63(7):894-909. doi: 10.1016/j.gie.2006.03.918. No abstract available. PMID 16733101
- [Result] Wu KL, Rayner CK, Chuah SK, Chiu KW, Lu CC, Chiu YC. Impact of low-residue diet on bowel preparation for colonoscopy. Dis Colon Rectum. 2011 Jan;54(1):107-12. doi: 10.1007/DCR.0b013e3181fb1e52. PMID 21160321
- [Result] Xie Q, Chen L, Zhao F, Zhou X, Huang P, Zhang L, Zhou D, Wei J, Wang W, Zheng S. A meta-analysis of randomized controlled trials of low-volume polyethylene glycol plus ascorbic acid versus standard-volume polyethylene glycol solution as bowel preparations for colonoscopy. PLoS One. 2014 Jun 5;9(6):e99092. doi: 10.1371/journal.pone.0099092. eCollection 2014. PMID 24902028
- [Derived] Barkun AN, Martel M, Epstein IL, Halle P, Hilsden RJ, James PD, Rostom A, Sey M, Singh H, Sultanian R, Telford JJ, von Renteln D. The Bowel CLEANsing National Initiative: High-Volume Split-Dose Vs Low-Volume Split-Dose Polyethylene Glycol Preparations: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1469-e1477. doi: 10.1016/j.cgh.2021.09.005. Epub 2021 Sep 9. PMID 34509641